CLINICAL TRIAL: NCT04547049
Title: An Open, Multi-center, Randomized Trial Comparing Haploidentical HSCTs From Young Non-first-degree and Older First-degree Donors in Hematological Malignancies
Brief Title: A Study Comparing Haploidentical Hematopoietic Stem Cell Transplantations (HSCTs) From Young Non-first-degree and Older First-degree Donors in Hematological Malignancies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yi Luo, Clinical Professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFD-001
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Leukemia
Keywords: hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia | interventions — Cytarabine; Busulfan; Cyclophosphamide; Semustine; thymoglobulin; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-first-degree donor (Active Comparator): Each patient receive graft from a non-first degree donor aged ≤40
  Conditoning regimens are decided by each center accoding to disease risk, patient age & status, and cormobidity index.The centers are required to use the same principle when treating NFD and FD patients. The used protocol in the current study included:
  For MAC: use BU-CY-based (described in detail)
  For RIC: use BUFlu:
  Drug: Fludarabine 30 mg/m²/kg, administered IV d-10 through d-5. Drug: Busulfan, 3.2 mg/kg/day administered IV day -6 (BU2) or -7 through -5 (BU3).
  Other conditioning regimen may include:
  FluMel, TBF, FTM, Cy-TBI, Flu-TBI.
  Interventions: Drug: Cytarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Me-CCNU; Drug: Rabbit antithymocyte globulin; Procedure: Allogeneic HSCT; Drug: Cyclosporin A; Drug: Mycophenolate Mofetil; Drug: MTX
- First-degree donor (Active Comparator): Each patients receive graft from a first-degree donor aged >50
  Conditoning regimens are decided by each center accoding to disease risk, patient age & status, and cormobidity index.The centers are required to use the same principle when treating NFD and FD patients. The used protocol in the current study included: For MAC: use BU-CY-based (described in detail) For RIC: use BUFlu: Drug: Fludarabine 30 mg/m²/kg, administered IV d-10 through d-5. Drug: Busulfan, 3.2 mg/kg/day administered IV day -6 (BU2) or -7 through -5 (BU3). Other conditioning regimen may include: FluMel, TBF, FTM, Cy-TBI, Flu-TBI.
  Interventions: Drug: Cytarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Me-CCNU; Drug: Rabbit antithymocyte globulin; Procedure: Allogeneic HSCT; Drug: Cyclosporin A; Drug: Mycophenolate Mofetil; Drug: MTX

INTERVENTIONS:
Drug: Cytarabine — 4 mg/m2/day administered IV day -10 through -9.
Drug: Busulfan — 3.2 mg/kg/day administered IV day -8 through -6.
Drug: Cyclophosphamide — 1.8 g/m2/day administered IV day -5 through -4.
Drug: Me-CCNU — 250mg/m2 once administered orally on day -3.
Drug: Rabbit antithymocyte globulin — Between 6mg/kg total dose administered IV day -5 through -2 AND 7.5mg/kg total dose administered IV day -5 through -2.
Procedure: Allogeneic HSCT — Day 0
Drug: Cyclosporin A — 2.5 mg/kg/day administered intravenously from day -7, target: 200-300ng/mL. Usually tapered during the second month, and ended in complete withdrawal during the ninth month after transplantation.
Drug: Mycophenolate Mofetil — 500 mg/day administered intravenously from day -9, ended in complete withdrawal on day +100.
Drug: MTX — 15 mg/m2 administered intravenously on day +1, 10mg/m2 on day +3, +6, and +9.

SUMMARY:
An open, multi-center, randomized trial comparing haploidentical HSCTs from young non-first-degree and older first-degree donors in hematological malignancies

DETAILED DESCRIPTION:
This is an open, multi-center, randomized trial comparing the clinical outcomes of haploidentical HSCTs from young non-first-degree and older first-degree donors in hematological malignancies. This study is indicated for patients with hematological malignancies including acute leukemias and MDS who are eligible to haploidentical HSCTs. 2 groups of patients will be enrolled with 88 in each group. The clinical criteria including survival, relapse, transplantation-related mortality will be monitored.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient age 13-78 years
* Absence of a suitable HLA identical related or unrelated hematopoietic stem cell donor
* Absence of a suitable partially HLA-mismatched (haploidentical), first-degree related donor aged between 18 and 50
* Presence of both HLA haploidentical young non-first-degree (age ≤ 40) and older first-degree (age >50) donors

Eligible diagnoses:

AML（excluding APL） with at least one of the following:

* median- or high- risk according to the WHO prognostic stratification system
* failure to achieve CR after 2 cycles of induction chemotherapy
* AML arising from MDS or a myeloproliferative disorder, or secondary AML
* patients in CR2 or beyond

Mixed-phenotype acute leukemia (MPAL) in morphological remission Acute lymphoblastic leukemia (T or B) in morphological remission

MDS with at least one of the following:

* IPSS score of INT-2 or greater
* IPSS score of INT-1 with life-threatening cytopenias, including those generally requiring greater than weekly transfusions

  * A first allo-HCT
  * Adequate end-organ function
  * ECOG performance status < 2
  * No other contraindications for HSCT
  * Signature of the informed consent

Patient Exclusion Criteria

* Availability of suitable HLA identical related or unrelated hematopoietic stem cell donors
* Availability of suitable partially HLA-mismatched (haploidentical), first-degree related donor aged between 18 and 50
* Not the first allo-HCT
* Presence of uncontrolled bacterial, viral, or fungal infection
* Patients with severe heart, lung, liver and kidney insufficiency
* HIV-positive patients
* Women of childbearing potential who are pregnant (β-HCG+) or breast feeding
* Patients with a psychiatric history
* ECOG performance status ≥ 3
* Patients with malignancies other than the primary disease
* Refusal to sign the informed consent

Donor Inclusion Criteria:

* The donor and recipient must be HLA haploidentical
* Meets institutional selection criteria and medically fit to donate
* Lack of recipient anti-donor HLA antibody

Donor Exclusion Criteria:

* The donor and recipient are HLA identical
* Has not donated blood products to recipient

Ages: 13 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of transplant-related nonrelapse mortality (NRM) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Progression-free survival (PFS) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of disease relapse or progression | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
GVHD-free, relapse-free survival (GRFS) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
  GRFS is defined as survival with no evidence of relapse/progression, grade III to IV aGVHD, and systemic therapy-requiring cGVHD.
Cumulative incidence of acute grade II-IV GVHD | 180 days
  Date of symptom onset, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of grade II or higher acute GVHD and grade III-IV acute GVHD will be recorded.
Cumulative incidence of chronic GVHD | 2 years
  Date of symptom onset, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of chronic GVHD and severe chronic GVHD will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - Xiangya Hospital Central South University, Changsha
  - Xinqiao Hospital, State Key Laboratory of Trauma and Chemical Poisoning, Army Medical University, Chongqing
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - The Affiliated People's Hospital of Ningbo University, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The First Affiliated Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No